CLINICAL TRIAL: NCT04910022
Title: A Phase I/II Combination Study of NMS-03305293 and Temozolomide in Adult Patients With Recurrent Glioblastoma
Brief Title: Ph I/II Study of NMS-03305293+TMZ in Adult Patients With Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PARPA-293-002; 2020-003417-35 (EudraCT Number); 2023-508318-41-00 (EU CTIS Number)
Record Dates: First submitted 2021-05-21; First posted 2021-06-02 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Diffuse Glioma
Keywords: IDH wild type; PARP inhibitor
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NMS-03305293 +TMZ (Experimental): Phase 1 Dose Escalation: All patients will receive NMS-03305293 and temozolomide (TMZ) administered orally (NMS-03305293 once or twice daily on days 1-7 or 28 consecutive days from Day 1 to Day 28; TMZ once daily on days 1-5;) in repeated 4-week cycles aimed at defining the Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Doses (RP2Ds) of NMS-03305293 in combination with TMZ. Each cycle is 28 days.
  Phase 2: Once the RP2D is defined, the patients will receive TMZ daily on days 1-5 in combination with NMS-03305293 at the RP2D on days 1-7 or on days 1-28 every 28 days.
  Backfill cohorts: additional patients may be treated with TMZ daily on days 1-5 and NMS-03305293 at different dose levels/schedules that have been previously assessed and determined to be safe, in order to properly characterize the exposure relationship over a range of doses/schedules. The backfill cohorts may run in parallel.
  Interventions: Drug: NMS-03305293; Drug: Temozolomide

INTERVENTIONS:
Drug: NMS-03305293 — Route of administration: Oral
Drug: Temozolomide — Route of administration: Oral
  Commercially available temozolomide

SUMMARY:
Multicenter, open-label, single-arm Phase 1/2 study on the safety and efficacy of the combination of NMS-03305293 and temozolomide (TMZ) in adult patients with diffuse gliomas (Phase 1) and isocitrate dehydrogenase (IDH) wild type glioblastoma (Phase 2) at first relapse.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1

  1. Histologically confirmed diagnosis of an intracranial diffuse glioma (i.e. diffuse astrocytoma, oligodendroglioma or glioblastoma). Sponsor may opt to restrict enrollment based on MGMT status, tumor type, tumor measurability or apply restriction on time to first relapse.
  2. Patients at first radiographic relapse after chemotherapy including temozolomide as long as no more than 12 cycles of temozolomide were administered.
  3. Patients may have been operated for recurrence. If operated:

     * residual and measurable disease after surgery is not required but pathology must have confirmed tumor recurrence.
     * a post-surgery MRI should be available within 48 hours following surgery.
     * surgery completed at least 2 weeks before enrolment and patient clinical status should not be worsened respect to pre-surgery condition
* Backfill cohorts

  1. Histologically confirmed diagnosis of Glioblastoma, IDH-wildtype as per WHO 2021 classification, including IDH-wildtype diffuse and astrocytic glioma in adults if there is microvascular proliferation or necrosis or TERT promoter mutation or EGFR gene amplification or +7/-10 chromosome copy number changes or c-IMPACT-NOW 3 definition including diffuse astrocytic glioma, IDH-wildtype, with molecular features of glioblastoma, WHO Grade 4. IDH1 status must be assessed locally by immunohistochemistry (IHC). If IHC is performed and is negative, and patient is < 55 years old, sequencing or a PCR-based validated test must be performed to exclude other IDH1 or IDH2 most frequent mutations. Sponsor may opt to restrict enrollment based on MGMT status or apply restriction on time to first relapse.
  2. Patients must have measurable disease and meet standard of care resection, if indicated, and irradiation, if indicated, with concomitant temozolomide plus up to 6 cycles of adjuvant temozolomide consistent with local standards of care.
  3. Patients may have been operated for recurrence. If operated:

     * residual and measurable disease after surgery is required
     * a post-surgery MRI should be available within 48 hours following surgery
     * surgery completed at least 2 weeks before enrolment and patient clinical status should not be worsened respect to pre-surgery condition.
* Phase 2

  1. Histologically confirmed diagnosis of Glioblastoma, IDH-wildtype as per WHO 2021 classification, including IDH-wildtype diffuse and astrocytic glioma in adults if there is microvascular proliferation or necrosis or TERT promoter mutation or EGFR gene amplification or +7/-10 chromosome copy number changes or c-IMPACTNOW 3 definition including diffuse astrocytic glioma, IDH-wildtype, with molecular features of glioblastoma, WHO Grade 4. IDH1 status must be assessed locally by immunohistochemistry (IHC). If IHC is performed and is negative, and patient is < 55 years old, sequencing or a PCR-based validated test must be performed to exclude other IDH1 or IDH2 most frequent mutations. Sponsor may opt to restrict enrollment based on MGMT status or apply restriction on time to first relapse.
  2. Patients must have measurable disease at first radiographic relapse after initial standard therapy including temozolomide as long as no more than 6 cycles of adjuvant temozolomide were administered and provided that patient completed standard of care concurrent temozolomide and the radiation therapy; multiple surgeries are allowed as long as patient is at first relapse and TMZ was administered as standard of care.
  3. Patients may have been operated for recurrence. If operated:

     * residual and measurable disease after surgery is required
     * a post-surgery MRI should be available within 48 hours following surgery
     * surgery completed at least 2 weeks before enrolment and patient clinical status should not be worsened respect to pre-surgery condition.
* Phase 1 (including backfill) and Phase 2

  4. For non-operated patients with measurable disease in Phase I, for backfill and for all patients in Phase 2, recurrent disease must be defined by at least one bidimensionally measurable contrast-enhancing lesion with clearly defined margins with minimal diameters of 10 mm, visible on 2 or more axial slices 5 mm apart, based on MRI scan done within two weeks prior to enrolment.

  5. Patients on steroids should have stable or decreasing dose of steroids for 7 days prior to the baseline MRI scan.

  6. Life expectancy of at least 3 months.

  7. Able to undergo brain MRI scans with IV gadolinium.

  8. No evidence of symptomatic and acute intratumoral hemorrhage on MRI. Patients with MRI demonstrating old hemorrhage or subacute blood after a neurosurgical procedure (biopsy or resection) are eligible.

  9. Sufficient tissue representative of the disease available for central MGMT promoter methylation status (Phase I and II) and IDH status evaluation (Phase I).

  10. Male or female patients with age ≥ 18 years.

  11. ECOG performance status ≤2.

  12. Signed and dated IEC or IRB-approved Informed Consent.

  13. Resolution of all acute toxic effects (excluding alopecia) of any prior anticancer therapy to NCI CTCAE (Version 5.0) Grade ≤ 1 or to the baseline laboratory values as defined in Inclusion Criterion Number 14.

  14. Baseline laboratory values fulfilling the requirements declared into the Protocol

  15. Patients must use highly effective contraception or true abstinence. Female patients of childbearing potential must agree to use effective contraception or abstinence during the period of therapy and in the following 6 months plus 5x NMS-03305293 half-life (3 days) after discontinuation of study treatment. Being NMS-03305293 a potential CYP3A perpetrator, hormonal contraception may lose efficacy while on treatment with NMS-03305293, therefore this should be taken into account. Male patients must be surgically sterile or must agree to use highly effective contraception or true abstinence during the period of therapy and in the following 90 days plus 5x NMS-03305293 half-life (3 days) after discontinuation of study treatment.

  16. Ability to swallow capsules intact (without chewing, crushing, or opening).

  17. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study indications or procedures.

Exclusion Criteria:

1. Current enrollment in another interventional clinical trial.
2. Current treatment with other anticancer agents or devices, or treatment at recurrence with carmustine wafer implants and proteasome inhibitors.
3. Previous treatment with PCV (procarbazine, lomustine and vincristine) or any of its components, carmustine wafer implants, or bevacizumab.
4. Previous treatment with PARP inhibitors.
5. Major surgery, other than surgery for recurrent diffuse glioma, within 4 weeks prior to treatment.
6. Standard radiotherapy within the three months (12 weeks) prior to the diagnosis of progression unless the progression is clearly outside the radiation field (eg, beyond the high-dose region or 80% isodose line) or unless the recurrence is histologically proven.
7. Prior radiotherapy with a dose over 65 Gy, stereotactic radiosurgery or brachytherapy, unless the recurrence is histologically proven.
8. Use of full-dose anticoagulants unless the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks before enrollment
9. Treatment with concomitant medications known to be sensitive substrates of CYP2D6 and CYP2C19 that cannot be replaced with another treatment.
10. Treatment with enzyme-inducing anti-epileptic drugs (EIAED). Patients may be on non-EIAED or not be taking any anti-epileptic drugs. Patients previously on EIAED must be fully switched to non-EIAED at least 2 weeks prior to enrolment.
11. Pregnant or breast-feeding women.
12. Known hypersensitivity to any component of NMS-03305293 or TMZ drug formulations.
13. Known active infections (bacterial, fungal, viral including HIV positivity) requiring systemic treatment.
14. Patients with QTc interval ≥460 milliseconds for women, ≥450 milliseconds for men or with risk factors for torsade de pointes (e.g., uncontrolled heart failure, uncontrolled hypokalemia, history of prolonged QTc interval or family history of long QT syndrome). For patients receiving treatment with concomitant medications known to prolong the QTc interval, replacement with another treatment prior to enrollment is mandatory. If concomitant use of anti-emetics is considered essential for the care of the patients, instruction in protocol will be followed.
15. Active gastrointestinal disease (e.g., documented gastrointestinal ulcer, Crohn's disease, ulcerative colitis, or short gut syndrome) or other syndromes that would impact on drug absorption.
16. Any of the following in the past 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, active bleeding disorder.
17. Prior invasive malignancy (except for non melanoma skin cancer, carcinoma in situ or localized cancer) unless the patient has been disease-free and off therapy for that disease for ≥ 3 years.
18. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-09-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with first-cycle dose limiting toxicity | Time interval between the first dose administration in Cycle 1 and the first dose administration in Cycle 2 which is expected to be 28 days or up to 42 days in case of dose delay due to drug related toxicity
Phase 2: Objective Response Rate | From the date of first response up to data cut-off (approximately 18 months)
  Objective Response Rate (ORR), calculated as the proportion of evaluable patients who have achieved, as best overall response (BOR), confirmed complete response (CR) or partial response (PR) through central retrospective assessment of RANO criteria

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From the Informed Consent signature to 28 days after the last dose of study treatment administration
  Safety will be assessed by adverse events (AEs), which include clinically significant abnormalities identified during a medical test (e.g. laboratory tests, electrocardiogram, vital signs, physical examinations). AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA) and their severity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).The analysis will focus on the events reported after the start of treatment (treatment emergent adverse events).
Maximum concentration (Cmax) of NMS-03305293 and possible identified metabolites (if appropriate) after single and multiple doses of drug | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Time to observed Cmax (Tmax) of NMS-03305293 and possible identified metabolites (if appropriate) after single and multiple doses of drug | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Area under the concentration-time curve up to the last detectable plasma concentration (AUClast) of NMS-03305293 and possible identified metabolites (if appropriate) after single and repeated dose of drug. | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Terminal elimination half-life (t1/2) of NMS-03305293 and possible identified metabolites (if appropriate) after single and multiple doses of drug | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Area under the plasma concentration vs. time curve to infinity (AUCinf) of NMS-03305293 and possible identified metabolites (if appropriate) after multiple doses of drug. | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Accumulation ratio (Rac) of NMS-03305293 and possible identified metabolites (if appropriate) after multiple doses of drug. | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Oral plasma clearance (CL/F) of NMS-03305293 and possible identified metabolites (if appropriate) after multiple doses of drug | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Apparent volume of distribution (Vd/F) of NMS-03305293 and possible identified metabolites (if appropriate) after multiple doses of drug | Phase 1 and backfill cohorts: Cycle 1 (each cycle is 28 days) on Days 1, 2, 5, 6 and 8; Cycle 2 on Days 5 and 15 (day 15 only if 28 days schedule). Phase 2: Cycle 1 (Days 1 and 5), Cycle 2 (Day 5) and Cycle 3 or Cycle 4 (Day 5)
  Plasma samples will be collected and used for pharmacokinetics assessments
Phase 1: Renal clearance of NMS-03305293 and possible identified metabolites (if appropriate) after multiple doses of drug | At baseline, at Cycle 1 (each cycle is 28 days) Day 5 at different timepoints
  Urine samples will be collected in patients treated in the phase 1 and in backfill cohorts and used for pharmacokinetics assessments
Phase 1: Cumulative amount recovered unchanged in the urine (Ae) of NMS-03305293 and possible identified metabolites (if appropriate) after multiple doses of drug | At baseline, at Cycle 1 (each cycle is 28 days) Day 5 at different timepoints
  Urine samples will be collected in patients treated in the phase 1 and in backfill cohorts and used for pharmacokinetics assessments
Phase 1: Cumulative amount recovered unchanged in the urine expressed as a fraction of administered dose (Ae%) of NMS-03305293 and possible identified metabolites (if appropriate) after multiple doses of drug | At baseline, at Cycle 1 (each cycle is 28 days) Day 5 at different timepoints.
  Urine samples will be collected in patients treated in the phase 1 and in backfill cohorts and used for pharmacokinetics assessments
Phase 1: Objective Tumor Response | At baseline, every 8 weeks until disease progression or start of a new anticancer therapy (approximately 18 months).
  Complete and partial responses will be assessed according to RANO criteria
Phase 1: Duration of Response | From the date of first response up to data cut-off (approximately 18 months).
  Duration of response will be calculated from the date of either first CR or PR until the date of documented progression for patients who achieved CR or PR. Patients who died without report of progression will be considered non-events and censored at their last disease-free assessment date
Phase 1: Progression Free Survival | From the date of treatment initiation up to data cut-off (approximately 18 months)
  Progression Free Survival will be calculated from the date of treatment initiation to the date of first documentation of disease progression, or death due to any cause, whichever occurs first
Phase 2: Duration of response (DoR) through central retrospective assessment of RANO criteria | From the date of first response up to data cut-off (approximately 18 months).
  Duration of response will be calculated from the date of either first CR or PR until the date of documented progression for patients who achieved CR or PR. Patients who died without report of progression will be considered non-events and censored at their last disease-free assessment date
Phase 2: Progression-free survival (PFS) | From the date of treatment initiation up to data cut-off (approximately 18 months)
  Progression Free Survival will be calculated from the date of treatment initiation to the date of first documentation of disease progression, or death due to any cause, whichever occurs first
Phase 2: 6-month PFS Rate | From date of treatment initiation until the date of first documentation of progression or death for any cause, whichever occurs first, assessed up to 6 months
  Percentage of patients progressive-free at 6 months from treatment initiation
Phase 2: 9 and 12-Months Overall Survival Rates | From the date of treatment initiation until the date of death from any cause, assessed up to 9 and 12 months.
  Percentage of patients alive at 9 and 12 months from treatment initiation.
Overall Survival | From the date of treatment initiation up to data cut-off (approximately 24 months)
  Overall Survival will be calculated from the date of treatment initiation to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (18):
- United States (11):
  - Mayo Clinic Hospital - Phoenix, Phoenix, Arizona
  - University of California Irvine Medical Center (UCIMC) - Chao Family Comprehensive Cancer Center, Orange, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, University Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Medical Center - First Hill Campus, Seattle, Washington
- Italy (4):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Istituto Clinico Humanitas, Rozzano
- Erasmus Medical Center, Rotterdam, Netherlands
- PanOncology Trials (Pan American Center for Oncology Trials, LLC), Rio Piedras, Puerto Rico
- University Hospital Zurich, Zurich, Switzerland